CLINICAL TRIAL: NCT06413966
Title: Comparison on Recurrence Rate of Pneumothorax Between Mesh and Apical Pleurectomy After Video-Assisted Thoracoscopic Blebectomy/Bullectomy for Primary Spontaneous Pneumothorax: A Randomized Controlled Trial (Pilot Study)
Brief Title: Study Compares Pneumothorax Recurrence: Absorbable Mesh vs. Pleurectomy in Primary Spontaneous Pneumothorax.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Apichat Tantraworasin, Associate Professor Doctor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUR-2566-0393
Record Dates: First submitted 2024-03-21; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Primary Spontaneous Pneumothorax
Keywords: Primary Spontaneous Pneumothorax; Video-assisted Thoracoscopic Surgery; Apical pleurectomy; Partially absorbable mesh coverage; Recurrence rate of pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * Participants (Double-blinded) and Assessor (nurse who will be assigned for collecting perioperative and postoperative results after surgery)
  * After obtaining informed consent and the patient's agreement to participate in the study, the patients will be allocated block sizes of four and computer-generated random numbers in sequential order within opaque envelopes that are sealed. The allocation process follows a 1:1 ratio.
  * Those sealed envelopes were kept by the researcher. On the day of operation, after video-assisted thoracoscopic blebectomy/bullectomy will be done, a randomized envelope will be opened by the scrub nurse to determine which additional method would be used between partially absorbable mesh and apical pleurectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially absorbable mesh coverage group (Experimental): - This group of patient will receive partially absorbable mesh coverage (ULTRAPRO size 15 x 15 cm, Ethicon) as an additional procedure after VATs to blebectomy/bullectomy.
  Interventions: Procedure: Partially absorbable mesh
- Apical pleurectomy group (Active Comparator): - This group of patient will receive standard surgical treatment that is used at Maharaj Nakorn Chiangmai Hospital, which is blebectomy or bullectomy with apical pleurectomy under video-assisted thoracoscopic approach
  Interventions: Procedure: Apical pleurectomy

INTERVENTIONS:
Procedure: Partially absorbable mesh — - In this group, after bullectomy or blebectomy, partially absorbable mesh (ULTRAPRO size 15 x 15 cm, Ethicon) will be prepared and inserted into the pleural cavity through one of the working ports and placed at the apical part of the thoracic cage (over the staple line) using fixation device (ProTack™ 5 mm fixation device, Medtronic).
  Arms: Partially absorbable mesh coverage group
Procedure: Apical pleurectomy — - In apical pleurectomy group, after bullectomy or blebectomy, the parietal surface from the apex to the fifth rib was dissected and abraded using a curved dissector with a diathermy scratch pad. Abrasion was done until a uniform aspect of bloody pleura was obtained.
  Arms: Apical pleurectomy group

SUMMARY:
This is a prospective, randomized controlled trial (pilot study) that aims to determine the incidence of post-operative recurrent pneumothorax within one-year timeframe after video-assisted thoracoscopic blebectomy/bullectomy with either apical pleurectomy or partially absorbable mesh, as well as to assess the efficacy in preventing post-operative recurrence pneumothorax. Patients, aged more than or equal 20-year-old, with the diagnosis of primary spontaneous pneumothorax, who require video-assisted thoracoscopic surgery at Maharaj Nakorn Chiangmai Hospital, Chiang Mai University, Chiang Mai, Thailand, will be enrolled into this study. The inform consent will be obtained before the enrollment. Patients will be randomized to two groups; Partially absorbable mesh coverage group (intervention group) and Apical pleurectomy group (control group).

DETAILED DESCRIPTION:
Background/Literature Review:

Primary spontaneous pneumothorax (PSP) is one of the most common respiratory conditions that usually occurs in young patients. While not a serious illness, it is worrisome because of its high rate of recurrence, ranging from 17 to 54%. Initial management for PSP is pleural drainage by aspiration of chest tube thoracostomy. Surgical intervention is needed if there was persistent air leakage (more than or equal to 5 days) after chest tube insertion or recurrent pneumothorax.

According to the British Thoracic Surgery (BTS) guideline for spontaneous pneumothorax, both open thoracotomy and video-assisted thoracotomy to blebectomy with apical pleurectomy is comparable in treating difficult or recurrent pneumothorax and considered a mainstay of treatment. Video-assisted thoracoscopic surgery (VAT) is a preferred surgical method for treating recurrence PSP because of its minimal invasiveness and low morbidity, which includes shorter length of hospital stays, less post-operative pain and post-operative pulmonary dysfunction. However, the frequency of post-operative recurrent pneumothorax following VAT procedure is higher than that of a conventional open thoracotomy, with reports of less than 1 percent. This frequency for that of VAT ranges from 9.5 percent to 24.5 percent. Therefore, when employing a less invasive approach, this needs to be balanced against the slight increase in recurrence rate.

The possible risk factors for recurrent pneumothorax after VAT include staple line leakage, overlooked or concealed blebs, bullae degeneration, incomplete resection of blebs, emphysematous changes in the resected area and visceral pleura damage during procedures6. To minimize postoperative recurrence, other preventive measures were introduced in addition to apical pleurectomy, such as chemical8,9 and mechanical pleurodesis, fibrin glue, mesh covering, or a combination of these measures (e.g., fibrin glue with mesh coverage). However, aside from apical pleurectomy, which have been mentioned in the BTS guideline, there is currently no other conclusive additional procedure that has been considered as part of standard treatment, necessitating further research.

Chemical pleurodesis yields an excellent rate of success in minimizing postoperative recurrent pneumothorax. It is simple and considered a cost-effective method. However, complete pleural symphysis can impair a patient's pulmonary function and sometimes produce chronic chest pain. Pleurectomy also increases the risk of postoperative bleeding, resulting in a longer period of chest tube insertion and fibrothorax, which could be challenging for future thoracic surgery.

Apical pleurectomy is one of the most widely used procedures because of its safety and feasibility. It results in adhesion between the visceral and parietal pleura, preventing the recurrence of postoperative pneumothorax. According to systemic review, mechanical apical pleurectomy exhibits comparable results in terms of 1-year postoperative recurrence pneumothorax as apical pleurectomy after thoracoscopic stapled blebectomy/bullectomy (p-value of 0.821). However, it produces less residual chest pain and a lower rate of hemothorax than apical pleurectomy.

Mesh coverage is increasing in popularity due to its reduction in postoperative recurrent pneumothorax, postoperative bleeding, and postoperative pain16, comparing to other additive procedure, including apical pleurectomy. Despite of the fact that both apical pleurectomy and mesh coverage have a comparable result in preventing post-operative recurrent pneumothorax, patients who underwent mechanical apical pleurectomy experienced with more severe residual pain than those with mesh coverage. Previous study found that the use of absorbable mesh for staple line coverage after blebectomy/bullectomy can significantly decrease postoperative pneumothorax with a recurrence rate of 2.6%, compared with 9.5% in patients who received VATS after blebectomy/bullectomy alone. The previous studies also display similar surgical outcomes.

Additional mechanical pleurodesis after covering the staple line with absorbable cellulose mesh and fibrin glue can also significantly lower the recurrent rate of postoperative pneumothorax, with a recurrence rate of 4.0%.

The postoperative 1-year recurrence rate was 9.5% in the absorbable mesh with fibrin glue group and 10.7% in the mechanical pleurodesis group.

As demonstrated in the preceding paragraphs, mesh coverage, with or without additional techniques such as fibrin glue, has been utilized in numerous prospective and retrospective studies to reinforce visceral pleura and symphyseal effects in order to prevent post-operative recurrent pneumothorax. However, due to its limited application in Thai clinical practice, information regarding the effectiveness of this surgical technique in preventing post-operative recurrent pneumothorax is scarce. Therefore, our goal is to conduct a prospective randomized controlled trial (pilot study) to determine whether the use of mesh as an additional procedure is more effective than the conventional technique, which is apical pleurectomy, in terms of preventing post-operative recurrent pneumothorax in patients with PSP who underwent video-assisted thoracoscopic blebectomy/bullectomy.

Rationale:

In standard of care for patients diagnosed with PSP who met the criteria for surgical treatment at Maharaj Nakorn Chiangmai Hospital, blebectomy or bullectomy with apical pleurectomy under video-assisted thoracoscopic approach will be performed. The utilization of mesh coverage as a preventive measure remains uncommon in Maharaj Nakorn Chiangmai Hospital, as well as in the majority of hospitals throughout Thailand. This stands in contrast to Japan, Korea, or Taiwan, where the use of mesh coverage to prevent post-operative pneumothorax has produced favorable results. As a result, compared to the standard of care, which is apical pleurectomy, there are still not many studies done in Thailand to assess the efficacy of mesh in preventing postoperative pneumothorax. Therefore, the researcher is motivated to carry out this study in order to assess the efficacy of mesh. As of yet, the mesh remains incapable of distributing funds in accordance with the patient's healthcare coverage. As a result, funding requests are required to carry out this research investigation. Should the results prove to be significant, it could subsequently be implemented as an alternative or even become a standard treatment for patients with PSP who were surgical candidates at Maharaj Nakorn Chiangmai hospital. Furthermore, funds for this treatment, which includes the cost of the mesh, could possibly be deducted from the patients' healthcare coverage.

Objectives:

* Determine the incidence of post-operative recurrent pneumothorax within one-year timeframe after video-assisted thoracoscopic blebectomy/bullectomy with either apical pleurectomy or partially absorbable mesh.
* Assess the efficacy in preventing post-operative recurrence pneumothorax after video-assisted thoracoscopic blebectomy/bullectomy with either apical pleurectomy or partially absorbable mesh.
* To compare the peri-operative and post-operative outcomes, as well as post-operative complications, of these two surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients (both sex) with first or second episode of primary spontaneous pneumothorax (either ipsilateral or contralateral) who have meet at least one of the following criteria for surgery below.
* Persistent air leakage five days following the insertion of a chest tube to treat spontaneous pneumothorax3,26 or failure of lung re-expansion2
* Air leakage after surgery will be categorized into 4 grades based on Robert David Cerfolio Classification System27; Grade1 inspire and expire air leakage (continuous air leakage), Grade 2 inspire air leakage, Grade 3 expire air leakage and Grade 4 forced expire air leakage.
* No matter grade of air leakage, once patients have any grade of air leakage of 4-5 days after chest drain insertion, they will be diagnosed with persistent air leakage.
* Hemopneumothorax
* Bilateral pneumothorax
* Visible blebs on the initial plain chest film or computed tomography
* Professions at risk (Aircraft personals, divers)
* Aged more than or equal to 20 years old.

Exclusion Criteria:

* Hemothorax or Pneumothorax that requires bilateral thoracic surgery.
* Previous ipsilateral thoracic operation
* Other serious concomitant illnesses or medical conditions e.g., Congestive heart failure, unstable angina, history of myocardial infarction within 1 year prior to entering this study.
* History of significant neurologic or psychiatric disorder

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of pneumothorax after operation | From date of surgery until the date of last follow-up, assessed at least 12 months and up to 24 months
  Recurrence rate of ipsilateral pneumothorax at least one- year follow-up period and up to 24 months after video-assisted thoracoscopic bullectomy with either partially absorbable mesh or apical pleurectomy. Gold standard for detecting recurrent pneumothorax is chest radiography and it is defined as the presence of an ipsilateral pneumothorax of any size in the follow-up chest radiography.

SECONDARY OUTCOMES:
Operative time (minute) | From time of skin incision until time of skin closure during intraoperative period
  Time between skin incision to surgical wound closure, report in minutes
Postoperative chest tube duration (days) | From date of first postoperative day until the date of chest drain removal, assessed up to 30 days
  Duration of chest tube insertion
Postoperative pain (pain score) | From time of immediate postoperative period until time of the patient has been discharged or date of death from any cause, whichever came first, assessed up to 30 days
  Using Visual analog scale (scale range from 0-10)
Composite postoperative complications | From time of immediate postoperative until time of the patient has been discharged or date of death from any cause, whichever came first, assessed up to 30 days.
  composite postoperative complications include persistent air leaks (more than or equal to 5 days) after operation, Fever, Empyema, and Pneumonia
Hospitalization cost (baht) | From the date that patient has been admitted until the date that patient has been discharged or date of death from any cause during admitted, assessed up to 30 days
  Cost during hospitalization
Postoperative pleural effusion (ml) | From date of 1st postoperative day until date of chest drain removed, assessed up to 30 days
  The amount of pleural fluid per day until it has been removed.
Intraoperative blood loss (ml) | From time of skin incision until time of skin closure during operative period
  Blood loss collected by anesthesiologist or surgeon
Dosage of morphine use after postoperative period till discharged. | From time of immediate postoperative period until time of patient discharged from hospital, assessed up to 30 days
  The dosage of morphine using will be counted from immediate postoperative period till discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Apichat Tantraworasin, M.D, Ph.D., Principal Investigator — Chiang Mai University
Locations (1):
- Department of surgery, Faculty of medicine, Chiang Mai University Hospital, Chiang Mai, Chaing Mai, Thailand